CLINICAL TRIAL: NCT05466487
Title: Transcranial Alternating Stimulation in Rehabilitation: a Randomized Controlled Trial in Chronic Stroke Patients With Visuospatial Neglect
Brief Title: Non-Invasive Brain Stimulation as an Innovative Treatment for Chronic Neglect Patients
Acronym: NibsNeglect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL70256.068.19
Record Dates: First submitted 2022-07-18; First posted 2022-07-20 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Spatial Neglect
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tACS (Experimental)
  Interventions: Device: Transcranial Alternating Current Stimulation (tACS); Behavioral: Visual Scanning Training (VST)
- Sham tACS (Sham Comparator)
  Interventions: Device: Transcranial Alternating Current Stimulation (tACS); Behavioral: Visual Scanning Training (VST)

INTERVENTIONS:
Device: Transcranial Alternating Current Stimulation (tACS) — Stimulation frequency and peak-to-peak intensity will be set to 10Hz and 1.5 milliampere (mA), phase offset will be set to 0 and 100 cycles will be used for ramping up. At the start of the neglect training session, the tACS will be started. When the neglect training session is finished, after maximally 40 minutes, the tACS will be switched off.
Behavioral: Visual Scanning Training (VST) — The most common treatment for neglect is VST, which is an intensive compensation training (see Dutch guidelines for rehabilitation of neglect: Ten Brink, Van Kessel, & Nijboer, 2017). The aim of this training is to improve visual scanning behavior, that is, to encourage neglect patients to actively and consciously pay attention to stimuli on the contralesional side.

SUMMARY:
Background Stroke is a leading cause of neurological impairments in language, motor and cognitive functions. Next to traditional stroke treatment, Non-Invasive Brain Stimulation (NIBS) offers the potential to facilitate stroke recovery as a complementary approach. Here, we aim at exploiting the principles of NIBS, specifically transcranial Alternating Current Stimulation (tACS), to promote functional recovery of people with neglect symptoms following stroke.

Objective To determine whether neglect training complemented with tACS treatment in chronic stroke patients suffering from neglect improves neglect-related symptoms compared to neglect training with sham stimulation.

Study design Double-blind randomized placebo-controlled intervention study. After enrollment and completion of baseline measurements, participants are randomly assigned to either the active tACS group or sham (control) group.

Intervention We will combine an evidence based visual scanning training (VST) with 40 minutes of (active or sham) tACS at alpha frequency. The intervention is administered three times a week for a duration of six weeks.

Outcomes of the study Performance on standard, conventional neuropsychological tests, as well as on ADL observation scales.

ELIGIBILITY:
Inclusion Criteria:

* neurologically objectified stroke;
* stroke occurred when patient was 18-80 years of age;
* chronic stroke (>6 months post-stroke onset);
* sufficient comprehension and communication skills to benefit from training (based on clinical judgement); and
* a screening containing four neuropsychological tests will be performed to evaluate the current severity of the neglect, since the diagnosis of neglect may have been established months or even years ago in our sample of chronic stroke patients.

Exclusion Criteria:

* currently engaging in cognitive rehabilitation treatment or neglect treatment;
* physically or mentally unable to participate (based on clinical judgment);
* hemianopsia (based on clinical judgement);
* severe communicative disability, as task descriptions need to be understood;
* local scalp injuries*;
* eczema on scalp or psoriasis*;
* diagnosed (neuro)psychiatric or neurodegenerative diseases*;
* current alcohol and/or drug abuse*; and
* pregnancy*.

  * due to tACS safety considerations.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2023-03-24 (Actual); Study Completion 2023-03-24 (Actual)

PRIMARY OUTCOMES:
Star Cancellation Task | Testing will take place before the training (T0; baseline), after the first (T1), ninth (T2), and eighteenth (T3) training session, as well as one week (T4) and three months (T5) after termination of the training.
  Quality of search score

SECONDARY OUTCOMES:
Computerized Visual Detection Task | Testing will take place before the training (T0; baseline), after the first (T1), ninth (T2), and eighteenth (T3) training session, as well as one week (T4) and three months (T5) after termination of the training.
  Sum of weighted hits
McIntosh Line Bisection Task-digitized | Testing will take place before the training (T0; baseline), after the first (T1), ninth (T2), and eighteenth (T3) training session, as well as one week (T4) and three months (T5) after termination of the training.
  Endpoint weightings bias
Schenkenberg Line Bisection Task | Testing will take place before the training (T0; baseline), after the first (T1), ninth (T2), and eighteenth (T3) training session, as well as one week (T4) and three months (T5) after termination of the training.
  Relative deviation score
Baking Tray Task | Testing will take place before the training (T0; baseline), after the ninth (T2) training session, as well as one week (T4) and three months (T5) after termination of the training.
  Average x-coordinate
Catherine Bergego Scale | Testing will take place before the training (T0; baseline), after the ninth (T2) training session, as well as one week (T4) and three months (T5) after termination of the training.
  Total score. The CBS is a 10-item observation scale, and results in a total score of 0 (no neglect) to 30 (severe neglect).
Subjective Neglect Questionnaire | Testing will take place before the training (T0; baseline), after the ninth (T2) training session, as well as one week (T4) and three months (T5) after termination of the training.
  Total score. The SNQ is a 19-item questionnaire, and results in a total score of 19 (no reported problems) to 95 (many/frequently reported problems).

OTHER OUTCOMES:
EEG | Testing will take place before the training (T0; baseline), and after the eighteenth (T3) training session.
  Power of alpha frequency band

CONTACTS AND LOCATIONS:
Overall Officials: Alexander T. Sack, PhD, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Middag-van Spanje M, Nijboer TCW, Schepers J, van Heugten C, Sack AT, Schuhmann T. Alpha transcranial alternating current stimulation as add-on to neglect training: a randomized trial. Brain Commun. 2024 Aug 30;6(5):fcae287. doi: 10.1093/braincomms/fcae287. eCollection 2024. PMID 39301290
- [Derived] Middag-van Spanje M, Schuhmann T, Nijboer T, van der Werf O, Sack AT, van Heugten C. Study protocol of transcranial electrical stimulation at alpha frequency applied during rehabilitation: A randomized controlled trial in chronic stroke patients with visuospatial neglect. BMC Neurol. 2022 Nov 2;22(1):402. doi: 10.1186/s12883-022-02932-7. PMID 36324088